CLINICAL TRIAL: NCT00105235
Title: A Phase II Multicenter Trial to Assess the Safety and Efficacy of Campath-1H and Tacrolimus Followed By Immunosuppression Withdrawal in Liver Transplantation (ITN024ST)
Brief Title: Immune System Suppression With Alemtuzumab and Tacrolimus in Liver Transplantation Patients
Acronym: TILT
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: National Institute of Allergy and Infectious Diseases (NIAID) (NIH)
Collaborators: Immune Tolerance Network (ITN) (Network)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: DAIT ITN024ST
Record Dates: First submitted 2005-03-10; First posted 2005-03-11 (Estimated); Results first posted 2012-04-05 (Estimated); Last update posted 2012-12-27 (Estimated); Status verified 2012-11

CONDITIONS: Liver Disease; Liver Transplantation
Keywords: transplantation; liver transplant; rejection; tolerance; antibody induction
MeSH Terms: conditions — Liver Diseases; Rejection, Psychology | interventions — Alemtuzumab; Cyclosporine; Mycophenolic Acid; Tacrolimus; Liver Transplantation

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Alemtuzumab (Experimental): Liver transplant, with two in-patient infused doses of alemtuzumab; followed by maintenance immunotherapy with cyclosporine, mycophenolate mofetil, and/or tacrolimus; with possible immunosuppression withdrawal
  Interventions: Drug: Alemtuzumab; Drug: Cyclosporine; Drug: Mycophenolate mofetil; Drug: Tacrolimus; Procedure: Liver transplant; Procedure: Immunosuppression withdrawal

INTERVENTIONS:
Drug: Alemtuzumab — T-cell depleting monoclonal antibody; two doses by intravenous infusion on Days 0 and 4
  Other Names: Campath
Drug: Cyclosporine — Oral immunosuppressant
Drug: Mycophenolate mofetil — Oral immunosuppressant
  Other Names: CellCept
Drug: Tacrolimus — Oral immunosuppressant
  Other Names: FK-506; Fujimycin
Procedure: Liver transplant — Occurs at study entry
Procedure: Immunosuppression withdrawal — Beginning no earlier than Year 1

SUMMARY:
Alemtuzumab is a man-made antibody used to treat certain blood disorders. Tacrolimus is a drug used to decrease immune system activity in people who have received organ transplants so that the new organ will not be rejected. This study will determine whether treatment with alemtuzumab and tacrolimus is effective in preventing organ rejection and maintaining the recipient's health after liver transplantation in patients with end-stage liver disease, and whether gradual tapering of tacrolimus treatment is safe for these patients.

DETAILED DESCRIPTION:
Organ transplantation is a common procedure in hospitals, but organ rejection and serious side effects are potential problems for the patient. Alemtuzumab is a monoclonal antibody that binds to and depletes excess T cells in the bone marrow of leukemia patients. In this study, alemtuzumab will destroy the recipient's white blood cells (WBCs) at the time of transplantation. It is hoped that WBCs produced after alemtuzumab administration will recognize the transplanted liver as "self" and not reject the new liver.

Drugs that suppress the immune system, such as tacrolimus, have contributed to increased success of transplantation. However, to prevent organ rejection, transplant recipients need to take immunosuppressive drugs for the rest of their lives, and these drugs make patients more susceptible to infection, endangering their health and survival. Regimens that are less toxic to or can eventually be withdrawn from transplant recipients are needed. This study will evaluate the effects of two in-patient doses of alemtuzumab followed by maintenance antirejection medication given to liver transplant patients post-transplant. This study will also determine if post-transplant tacrolimus therapy can be slowly and safely tapered off and withdrawn a year after transplant. Participants in this study will be patients with end-stage liver disease who will undergo liver transplantation at the start of the study.

This study will last at least 2 years. Patients will undergo liver transplantation at the start of the study on Day 0. Patients will receive in-patient infusions of alemtuzumab on Days 0 and 4. Starting on Day 1, patients will receive oral cyclosporine, mycophenolate mofetil, and/or tacrolimus daily. Patients will be hospitalized for at least 1 week after transplantation. Because of suppression of patients' immune systems by alemtuzumab and these other immunosuppressants, they will also receive prophylactic medications for a minimum of 3 months after transplantation to prevent opportunistic infections.

There will be at least eight study visits; they will occur at Days 4, 7, and 14 and at Months 1, 3, 6, 9, and 12. Patients will have liver biopsies at Day 0 and Months 6 and 12. At Month 12, participants will have assessments and blood tests to determine if they meet certain criteria and are eligible to undergo tacrolimus tapering. Patients eligible for tapering will undergo a 12-month gradual withdrawal of tacrolimus; they will be followed for an additional 2 years, with study visits at Months 18, 24, 30, and 36. Patients ineligible for tacrolimus tapering will continue taking their antirejection medication for the duration of the study; they will be followed for an additional year, with study visits at Months 18 and 24.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of nonimmune, nonviral, end-stage liver disease
* Need liver transplant
* Willing to use acceptable means of contraception for the duration of the study

Exclusion Criteria:

* Previous transplant
* Multiorgan transplant or living donor transplant
* Donor liver from a donor positive for antibody against hepatitis B core antigen or hepatitis C virus
* Donor liver from a non-heart-beating donor
* Liver failure due to autoimmune disease, such as autoimmune hepatitis, primary sclerosing cholangitis, or primary biliary cirrhosis
* Hepatitis B or C virus infection
* HIV infection
* Stage III or higher hepatocellular cancer based on pre-transplant imaging
* History of cancer. Patients with hepatocellular cancer, adequately treated in situ cervical carcinoma, or adequately treated basal or squamous cell carcinoma of skin are not excluded.
* Active systemic infection at the time of transplantation
* Clinically significant chronic renal, cardiovascular, or cerebrovascular disease
* Any investigational drug within 6 weeks of study entry
* Hypersensitivity to alemtuzumab or tacrolimus

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 27 (Actual)
Dates: Start 2005-06; Primary Completion 2007-03 (Actual); Study Completion 2011-03 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: J. Richard Thistlethwaite, MD, Principal Investigator — University of Chicago
Locations (9):
- United States (8):
  - University of California, San Francisco, San Francisco, California
  - University of Colorado, Denver, Colorado
  - University of Miami School of Medicine, Miami, Florida
  - University of Michigan, Ann Arbor, Michigan
  - Cleveland Clinic, Cleveland, Ohio
  - University of Pennsylvania, Philadelphia, Pennsylvania
  - Baylor University, Dallas, Texas
  - University of Wisconsin, Madison, Wisconsin
- University of Alberta, Edmonton, Alberta, Canada

REFERENCES:
- [Background] First MR. Tacrolimus based immunosuppression. J Nephrol. 2004 Nov-Dec;17 Suppl 8:S25-31. PMID 15599882
- [Background] Tryphonopoulos P, Madariaga JR, Kato T, Nishida S, Levi DM, Moon J, Selvaggi G, De Faria W, Regev A, Bejarano P, Khaled A, Safdar K, Esquenazi V, Weppler D, Yoshida H, Ruiz P, Miller J, Tzakis AG. The impact of Campath 1H induction in adult liver allotransplantation. Transplant Proc. 2005 Mar;37(2):1203-4. doi: 10.1016/j.transproceed.2004.12.157. PMID 15848669
- [Background] Tzakis AG, Tryphonopoulos P, Kato T, Nishida S, Levi DM, Madariaga JR, Gaynor JJ, De Faria W, Regev A, Esquenazi V, Weppler D, Ruiz P, Miller J. Preliminary experience with alemtuzumab (Campath-1H) and low-dose tacrolimus immunosuppression in adult liver transplantation. Transplantation. 2004 Apr 27;77(8):1209-14. doi: 10.1097/01.tp.0000116562.15920.43. PMID 15114087
- See also: Click here for the Immune Tolerance Network Web site — http://www.immunetolerance.org

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Recruitment details: Eight centers in the United States and one center in Canada enrolled 27 participants with end-stage liver disease who met entry criteria between February 2005 and May 2006.
Groups:
- Alemtuzumab: Recipients of a liver allograft for end-stage liver disease received a 30 mg IV dose of alemtuzumab on study days 0 and 4 (immunosuppressive induction). Beginning on study day 1, participants received tacrolimus orally (dose adjusted to yield trough blood levels of 5-12 ng/mL) with or without mycophenolate orally (<= 1.5g twice daily), at the discretion of the investigator. Six months post transplant, the tacrolimus dose was adjusted to yield trough blood levels of 5-10 ng/mL. Participants with significant toxicities related to tacrolimus were changed to cyclosporine (CsA), with the dose adjusted to maintain trough blood levels of 200-350 ng/mL during the first 3 months post transplant and 100-300 ng/mL from month 4 until CsA tapering was initiated. Maintenance immunosuppression was maintained for at least 12 months. At 12 months, participants were assessed for immune reconstitution and for the ability to undergo tapering and subsequent withdrawal of immunosuppression
Period: Overall Study
Arm/Group | Alemtuzumab
Started | 27
Completed | 20
Not Completed | 7
Not completed — Death | 4
Not completed — Physician Decision | 1
Not completed — Withdrawal by Subject | 2

BASELINE CHARACTERISTICS:
Arm/Group | Alemtuzumab
Number analyzed (Participants) | 27
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 25
  >=65 years | 2
Age Continuous [Mean (Standard Deviation); unit: years] | 52.5 (10.3)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 8
  Male | 19
Region of Enrollment [Number; unit: participants]
  United States | 26
  Canada | 1

OUTCOME MEASURES:

1. Primary Outcome: Proportion of Participants Who Have Graft Loss or Death
Description: Proportion of participants who had liver graft loss or who died within 1 year of undergoing transplantation. Note: Participants who discontinued treatment or terminated the study prior to 1 year post transplantation are considered treatment failures and are included in this measure.
Time Frame: Within 1 year of post-transplantation
Population: Safety Sample
Measure: Number; unit: Proportion of Participants
Arm/Group | Alemtuzumab
Number analyzed (Participants) | 27
Proportion of Participants | 0.22
Statistical Analysis 1: Comparison: Alemtuzumab; Test type: Superiority or Other; Exact Binomial Confidence Interval; Proportion = 0.22, 95% CI 2-sided [.086 to .423]

2. Secondary Outcome: Proportion of Participants Who Had Graft Loss or Death
Description: Proportion of participants who had liver graft loss or who died or terminated from the study within 2 years of initiating immunosuppression withdrawal
Time Frame: Within 2 years after initiation of immunosuppression withdrawal
Population: Participants who initiated immunosuppression withdrawal
Measure: Number; unit: Proportion of Participants
Arm/Group | Alemtuzumab
Number analyzed (Participants) | 10
Proportion of Participants | 0
Statistical Analysis 1: Comparison: Alemtuzumab; Test type: Superiority or Other; Exact Binomial Confidence Interval; Proportion = 0, 95% CI 2-sided [0 to 0.3]

3. Secondary Outcome: Number of Events: Immunosuppression-related Complications
Description: Certain events are associated with immunosuppression. This measure looks at post-transplant infection, post-transplant malignancies, post-transplant diabetes, and post-transplant renal failure. Immunosuppression withdrawal is intended to reduce these type of events. However, reduction in immunosuppression can lead to complications in liver and renal function, as measured by acute rejection, chronic rejection, and post-transplant renal failure. Lower numbers for any of these events indicates greater success with transplantation and immunosuppression withdrawal (where applicable)
Time Frame: From transplantation until study completion or participant termination (participants followed up to 60 months)
Population: Safety Sample
Measure: Number; unit: Events
Groups:
- Withdrawal Never Started; Completed Withdrawal and Remains Off Immunosuppression; Completed Withdrawal and Restarted Immunosuppression; Discontinued Immunosuppression Withdrawal: Recipients of a liver allograft for end-stage liver disease received a 30 mg IV dose of alemtuzumab on study days 0 and 4 (immunosuppressive induction). Beginning on study day 1, participants received tacrolimus orally (dose adjusted to yield trough blood levels of 5-12 ng/mL) with or without mycophenolate orally (<= 1.5g twice daily), at the discretion of the investigator. Six months post transplant, the tacrolimus dose was adjusted to yield trough blood levels of 5-10 ng/mL. Participants with significant toxicities related to tacrolimus were changed to cyclosporine (CsA), with the dose adjusted to maintain trough blood levels of 200-350 ng/mL during the first 3 months post transplant and 100-300 ng/mL from month 4 until CsA tapering was initiated. Maintenance immunosuppression was maintained for at least 12 months. At 12 months, participants were assessed for immune reconstitution and for the ability to undergo tapering and subsequent withdrawal of immunosuppression
Arm/Group | Withdrawal Never Started | Completed Withdrawal and Remains Off Immunosuppression | Completed Withdrawal and Restarted Immunosuppression | Discontinued Immunosuppression Withdrawal
Number analyzed (Participants) | 17 | 2 | 2 | 6
Events
  Acute Rejection | 6 | 0 | 0 | 0
  Chronic Rejection | 1 | 0 | 0 | 0
  Post-transplant Infection | 76 | 2 | 10 | 11
  Post-transplant Malignancies | 1 | 0 | 0 | 0
  Post-transplant Diabetes | 0 | 0 | 0 | 1
  Post-transplant Renal Failure | 11 | 0 | 2 | 1

4. Secondary Outcome: Proportion of Participants Successfully Withdrawn From Immunosuppressants
Description: This measure of tolerance induction includes the proportion of participants who qualify for immunosuppression withdrawal as determined by a review of individual clinical results by a protocol withdrawal committee. Successful withdrawal definition: participants who remain off immunosuppression for at least 8 weeks.
Time Frame: From 1 year post- transplantation until study completion or participant termination (participants followed up to 48 months post-transplant)
Population: Intent-to-treat
Measure: Number; unit: Proportion of Participants
Arm/Group | Alemtuzumab
Number analyzed (Participants) | 27
Proportion of Participants | 0.2
Statistical Analysis 1: Comparison: Alemtuzumab; Test type: Superiority or Other; Exact Binomial Confidence Interval; Proportion = 0.2, 95% CI 2-sided [0.04 to 0.3]

5. Secondary Outcome: Proportion of Participants Successfully Withdrawn and Remain Off Immunosuppressants
Description: This measure of tolerance induction includes the proportion of participants who qualify for immunosuppression withdrawal as determined by a review of individual clinical results by a protocol withdrawal committee, were successfully withdrawn from immunosuppressants, and remained off immunosuppressants at the time the trial ended. Successful withdrawal definition: participants who remain off immunosuppression for at least 8 weeks and do not restart immunosuppressant drugs after successful withdrawal.
Time Frame: as for outcome 4
Population: Intent-to-treat
Measure: Number; unit: Proportion of Participants
Arm/Group | Alemtuzumab
Number analyzed (Participants) | 27
Proportion of Participants | 0.1
Statistical Analysis 1: Comparison: Alemtuzumab; Test type: Superiority or Other; Exact Binomial Confidence Interval; Proportion = 0.1, 95% CI 2-sided [0.01 to 0.2]

ADVERSE EVENTS:
Time Frame: From transplantation until study completion or participant termination (participants followed up to 48 months post-transplantation)
Description: This study graded the severity of adverse events experienced by the study participant according to criteria set forth in the National Cancer Institute's Common Terminology Criteria for Adverse Events Version 3.0 (June 10, 2003)
Arm/Group | Alemtuzumab
Serious Adverse Events (participants affected / at risk) | 27/27
Other Adverse Events (participants affected / at risk) | 26/27
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Alemtuzumab (N=27)
Anaemia (Blood and lymphatic system disorders) | 3 (3)
Coagulopathy (Blood and lymphatic system disorders) | 1 (1)
Neutropenia (Blood and lymphatic system disorders) | 1 (1)
Pancytopenia (Blood and lymphatic system disorders) | 1 (1)
Thrombocytopenia (Blood and lymphatic system disorders) | 2 (2)
Bradycardia (Cardiac disorders) | 1 (1)
Cardio-respiratory arrest (Cardiac disorders) | 1 (1)
Tachycardia (Cardiac disorders) | 1 (1)
Ventricular tachycardia (Cardiac disorders) | 1 (1)
Abdominal discomfort (Gastrointestinal disorders) | 1 (1)
Ascites (Gastrointestinal disorders) | 1 (2)
Gastric ileus (Gastrointestinal disorders) | 1 (1)
Gastrointestinal haemorrhage (Gastrointestinal disorders) | 2 (2)
Oesophageal varices haemorrhage (Gastrointestinal disorders) | 1 (1)
Peritoneal haemorrhage (Gastrointestinal disorders) | 1 (1)
Umbilical hernia (Gastrointestinal disorders) | 1 (1)
Varices oesophageal (Gastrointestinal disorders) | 1 (1)
Chest pain (General disorders) | 1 (1)
Multi-organ failure (General disorders) | 1 (1)
Pyrexia (General disorders) | 2 (4)
Bile duct stenosis (Hepatobiliary disorders) | 6 (8)
Cholestasis (Hepatobiliary disorders) | 1 (1)
Hepatic artery thrombosis (Hepatobiliary disorders) | 1 (1)
Hepatic cirrhosis (Hepatobiliary disorders) | 1 (1)
Hepatic failure (Hepatobiliary disorders) | 1 (1)
Hepatic steatosis (Hepatobiliary disorders) | 2 (2)
Liver disorder (Hepatobiliary disorders) | 1 (1)
Hypersensitivity (Immune system disorders) | 1 (1)
Transplant rejection (Immune system disorders) | 9 (12)
Abdominal infection (Infections and infestations) | 1 (1)
Bacteraemia (Infections and infestations) | 2 (3)
Clostridium difficile colitis (Infections and infestations) | 1 (1)
Endocarditis (Infections and infestations) | 1 (1)
Gastroenteritis viral (Infections and infestations) | 1 (1)
Hydrocele male infected (Infections and infestations) | 1 (1)
Influenza (Infections and infestations) | 1 (1)
Liver abscess (Infections and infestations) | 1 (1)
Lung infection pseudomonal (Infections and infestations) | 2 (2)
Osteomyelitis (Infections and infestations) | 1 (1)
Peritonitis bacterial (Infections and infestations) | 3 (3)
Pneumonia (Infections and infestations) | 2 (2)
Sepsis (Infections and infestations) | 3 (4)
Urinary tract infection (Infections and infestations) | 2 (2)
Urinary tract infection enterococcal (Infections and infestations) | 1 (1)
Wound infection (Infections and infestations) | 1 (1)
Collapse of lung (Injury, poisoning and procedural complications) | 1 (1)
Femoral neck fracture (Injury, poisoning and procedural complications) | 1 (1)
Graft loss (Injury, poisoning and procedural complications) | 1 (1)
Hip fracture (Injury, poisoning and procedural complications) | 2 (2)
Post procedural haemorrhage (Injury, poisoning and procedural complications) | 2 (2)
Road traffic accident (Injury, poisoning and procedural complications) | 1 (1)
Venous injury (Injury, poisoning and procedural complications) | 1 (1)
Weaning failure (Injury, poisoning and procedural complications) | 1 (1)
Liver function test abnormal (Investigations) | 3 (3)
Dehydration (Metabolism and nutrition disorders) | 2 (3)
Hyperkalaemia (Metabolism and nutrition disorders) | 2 (3)
Hypoglycaemia (Metabolism and nutrition disorders) | 1 (1)
Metabolic acidosis (Metabolism and nutrition disorders) | 2 (2)
B-cell lymphoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1)
Benign small intestinal neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1)
Hepatic neoplasm malignant (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1)
Squamous cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1)
Central pontine myelinolysis (Nervous system disorders) | 1 (1)
Mental status changes (Psychiatric disorders) | 2 (2)
Paranoia (Psychiatric disorders) | 1 (1)
Renal failure (Renal and urinary disorders) | 1 (1)
Renal failure acute (Renal and urinary disorders) | 3 (3)
Renal tubular necrosis (Renal and urinary disorders) | 1 (1)
Menorrhagia (Reproductive system and breast disorders) | 1 (1)
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 4 (4)
Hypercapnia (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 2 (2)
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Respiratory arrest (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Respiratory distress (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Respiratory failure (Respiratory, thoracic and mediastinal disorders) | 3 (3)
Deep vein thrombosis (Vascular disorders) | 2 (2)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Alemtuzumab (N=27)
Anaemia (Blood and lymphatic system disorders) | 18 (36)
Coagulopathy (Blood and lymphatic system disorders) | 3 (4)
Leukopenia (Blood and lymphatic system disorders) | 10 (16)
Lymphopenia (Blood and lymphatic system disorders) | 2 (2)
Neutropenia (Blood and lymphatic system disorders) | 7 (9)
Splenomegaly (Blood and lymphatic system disorders) | 2 (2)
Thrombocytopenia (Blood and lymphatic system disorders) | 9 (16)
Atrial fibrillation (Cardiac disorders) | 2 (3)
Bradycardia (Cardiac disorders) | 2 (2)
Palpitations (Cardiac disorders) | 2 (2)
Pericardial effusion (Cardiac disorders) | 2 (3)
Tachycardia (Cardiac disorders) | 4 (4)
Ear pain (Ear and labyrinth disorders) | 2 (2)
Hypothyroidism (Endocrine disorders) | 4 (4)
Ocular icterus (Eye disorders) | 2 (2)
Abdominal discomfort (Gastrointestinal disorders) | 3 (3)
Abdominal distension (Gastrointestinal disorders) | 9 (13)
Abdominal pain (Gastrointestinal disorders) | 11 (16)
Abdominal pain upper (Gastrointestinal disorders) | 3 (3)
Ascites (Gastrointestinal disorders) | 5 (7)
Constipation (Gastrointestinal disorders) | 17 (30)
Diarrhoea (Gastrointestinal disorders) | 15 (23)
Diverticulum (Gastrointestinal disorders) | 2 (2)
Dyspepsia (Gastrointestinal disorders) | 5 (6)
Dysphagia (Gastrointestinal disorders) | 3 (3)
Flatulence (Gastrointestinal disorders) | 2 (2)
Ileus (Gastrointestinal disorders) | 2 (2)
Nausea (Gastrointestinal disorders) | 16 (24)
Umbilical hernia (Gastrointestinal disorders) | 2 (2)
Vomiting (Gastrointestinal disorders) | 5 (7)
Asthenia (General disorders) | 4 (4)
Fatigue (General disorders) | 4 (4)
Generalised oedema (General disorders) | 6 (7)
Oedema (General disorders) | 6 (8)
Oedema peripheral (General disorders) | 16 (24)
Pain (General disorders) | 11 (17)
Pyrexia (General disorders) | 13 (25)
Cholangitis (Hepatobiliary disorders) | 2 (2)
Cholestasis (Hepatobiliary disorders) | 6 (6)
Hepatic steatosis (Hepatobiliary disorders) | 4 (4)
Hyperbilirubinaemia (Hepatobiliary disorders) | 5 (5)
Jaundice (Hepatobiliary disorders) | 9 (11)
Bacteraemia (Infections and infestations) | 4 (6)
Cellulitis (Infections and infestations) | 2 (3)
Clostridium difficile colitis (Infections and infestations) | 3 (4)
Cytomegalovirus infection (Infections and infestations) | 2 (2)
Fungal skin infection (Infections and infestations) | 3 (3)
Localised infection (Infections and infestations) | 2 (2)
Peritoneal infection (Infections and infestations) | 2 (2)
Pneumonia (Infections and infestations) | 3 (3)
Sinusitis (Infections and infestations) | 2 (5)
Urinary tract infection (Infections and infestations) | 5 (8)
Wound infection (Infections and infestations) | 2 (3)
Endotracheal intubation complication (Injury, poisoning and procedural complications) | 2 (2)
Incision site pain (Injury, poisoning and procedural complications) | 7 (8)
Incisional hernia (Injury, poisoning and procedural complications) | 3 (4)
Operative haemorrhage (Injury, poisoning and procedural complications) | 2 (2)
Post procedural bile leak (Injury, poisoning and procedural complications) | 3 (4)
Post procedural haemorrhage (Injury, poisoning and procedural complications) | 2 (2)
Procedural complication (Injury, poisoning and procedural complications) | 2 (2)
Procedural hypotension (Injury, poisoning and procedural complications) | 2 (3)
Procedural pain (Injury, poisoning and procedural complications) | 8 (9)
Wound secretion (Injury, poisoning and procedural complications) | 2 (2)
Blood alkaline phosphatase increased (Investigations) | 3 (3)
Blood creatinine increased (Investigations) | 7 (15)
Blood magnesium decreased (Investigations) | 4 (7)
Blood phosphorus decreased (Investigations) | 2 (4)
Breath sounds abnormal (Investigations) | 4 (6)
Cardiac murmur (Investigations) | 5 (5)
Coagulation time prolonged (Investigations) | 2 (3)
Electrocardiogram abnormal (Investigations) | 2 (2)
Haematocrit decreased (Investigations) | 2 (2)
Hepatic enzyme increased (Investigations) | 2 (2)
International normalised ratio increased (Investigations) | 3 (3)
Liver function test abnormal (Investigations) | 8 (8)
Platelet count decreased (Investigations) | 3 (3)
Acidosis (Metabolism and nutrition disorders) | 2 (2)
Anorexia (Metabolism and nutrition disorders) | 4 (4)
Cachexia (Metabolism and nutrition disorders) | 3 (3)
Decreased appetite (Metabolism and nutrition disorders) | 5 (5)
Dehydration (Metabolism and nutrition disorders) | 7 (7)
Failure to thrive (Metabolism and nutrition disorders) | 2 (2)
Fluid overload (Metabolism and nutrition disorders) | 6 (8)
Hyperglycaemia (Metabolism and nutrition disorders) | 14 (19)
Hyperkalaemia (Metabolism and nutrition disorders) | 14 (24)
Hyperlipidaemia (Metabolism and nutrition disorders) | 2 (2)
Hyperphosphataemia (Metabolism and nutrition disorders) | 3 (3)
Hypoalbuminaemia (Metabolism and nutrition disorders) | 3 (3)
Hypocalcaemia (Metabolism and nutrition disorders) | 8 (8)
Hypoglycaemia (Metabolism and nutrition disorders) | 3 (4)
Hypokalaemia (Metabolism and nutrition disorders) | 14 (21)
Hypomagnesaemia (Metabolism and nutrition disorders) | 10 (19)
Hyponatraemia (Metabolism and nutrition disorders) | 5 (5)
Hypophosphataemia (Metabolism and nutrition disorders) | 2 (2)
Hypovolaemia (Metabolism and nutrition disorders) | 3 (4)
Metabolic acidosis (Metabolism and nutrition disorders) | 3 (4)
Metabolic alkalosis (Metabolism and nutrition disorders) | 2 (3)
Arthralgia (Musculoskeletal and connective tissue disorders) | 3 (3)
Back pain (Musculoskeletal and connective tissue disorders) | 8 (10)
Muscle atrophy (Musculoskeletal and connective tissue disorders) | 3 (3)
Muscle spasms (Musculoskeletal and connective tissue disorders) | 4 (4)
Musculoskeletal pain (Musculoskeletal and connective tissue disorders) | 2 (2)
Dizziness (Nervous system disorders) | 2 (2)
Dysarthria (Nervous system disorders) | 2 (2)
Headache (Nervous system disorders) | 9 (13)
Neurotoxicity (Nervous system disorders) | 2 (2)
Sciatica (Nervous system disorders) | 2 (2)
Tremor (Nervous system disorders) | 7 (9)
Agitation (Psychiatric disorders) | 6 (8)
Anxiety (Psychiatric disorders) | 7 (7)
Confusional state (Psychiatric disorders) | 5 (5)
Depression (Psychiatric disorders) | 7 (8)
Insomnia (Psychiatric disorders) | 15 (20)
Mental status changes (Psychiatric disorders) | 2 (2)
Renal failure (Renal and urinary disorders) | 7 (7)
Renal failure acute (Renal and urinary disorders) | 3 (3)
Scrotal oedema (Reproductive system and breast disorders) | 2 (3)
Atelectasis (Respiratory, thoracic and mediastinal disorders) | 6 (6)
Cough (Respiratory, thoracic and mediastinal disorders) | 5 (8)
Dysphonia (Respiratory, thoracic and mediastinal disorders) | 2 (2)
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 5 (7)
Nasal congestion (Respiratory, thoracic and mediastinal disorders) | 2 (2)
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 6 (7)
Pneumothorax (Respiratory, thoracic and mediastinal disorders) | 2 (2)
Productive cough (Respiratory, thoracic and mediastinal disorders) | 4 (4)
Pulmonary oedema (Respiratory, thoracic and mediastinal disorders) | 4 (5)
Rales (Respiratory, thoracic and mediastinal disorders) | 3 (3)
Tachypnoea (Respiratory, thoracic and mediastinal disorders) | 2 (2)
Wheezing (Respiratory, thoracic and mediastinal disorders) | 8 (8)
Ecchymosis (Skin and subcutaneous tissue disorders) | 2 (2)
Night sweats (Skin and subcutaneous tissue disorders) | 2 (2)
Petechiae (Skin and subcutaneous tissue disorders) | 2 (3)
Pruritus (Skin and subcutaneous tissue disorders) | 10 (12)
Rash (Skin and subcutaneous tissue disorders) | 5 (7)
Skin ulcer (Skin and subcutaneous tissue disorders) | 5 (5)
Urticaria (Skin and subcutaneous tissue disorders) | 2 (2)
Wound drainage (Surgical and medical procedures) | 2 (2)
Deep vein thrombosis (Vascular disorders) | 3 (3)
Haematoma (Vascular disorders) | 2 (2)
Haemorrhage (Vascular disorders) | 2 (2)
Hypertension (Vascular disorders) | 16 (17)
Hypotension (Vascular disorders) | 8 (15)

LIMITATIONS AND CAVEATS:
This study was converted to a pilot study on May 23, 2006. Only 27 of the planned 211 participants were enrolled, thus reducing the number of subjects available for analysis.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No